CLINICAL TRIAL: NCT07167290
Title: SCI-FACT: The Acceptability and Effectiveness of Delivering a Focused Acceptance and Commitment Therapy Intervention in Inpatient Spinal Cord Injury Rehabilitation Settings
Brief Title: SCI-FACT: The Effectiveness of Focused ACT for SCI Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25005
Record Dates: First submitted 2025-07-24; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Acceptance and Commitment Therapy; Brief Intervention
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A single case experimental design (SCED) series will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused Acceptance and Commitment Therapy (Experimental): All participants will be in this arm and will receive a focused acceptance and commitment therapy intervention. This will be delivered over 1-3 sessions and be based on the facilitators handbook that will be provided to clinicians.
  Interventions: Behavioral: Focused Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Focused Acceptance and Commitment Therapy — Focused Acceptance and Commitment Therapy will be delivered following a facilitators guide. The intervention is adapted for Spinal Cord Injury patients and is to be delivered on an inpatient neurorehabilitation setting over the course of 1-3 sessions.

SUMMARY:
Research has found that patients with a Spinal Cord Injury (SCI) suffer with longstanding mental health difficulties, likely due to the impact of the lifelong physical and health problems that come with their injury. Therefore, it is important to make sure that there is effective psychological support available to them. Unfortunately, research shows that the most commonly used therapy approach, CBT, has very inconsistent evidence regarding its effectiveness for SCI patients. It has also been found that providing support shortly after the injury can be helpful for patients in the long term. Therefore, this study aims to evaluate whether an alternative therapy approach, called Focused Acceptance and Commitment Therapy (FACT), can be effectively delivered to SCI patients shortly after their injury, whilst they are recovering in hospital.

To answer this question, a single case experimental design (SCED) series will be used in which participants will regularly complete a number of questionnaires asking about: symptoms relating to their mental health; quality of life; how they are adjusting to their injury; and how they approach coping with difficulties they face, before receiving FACT and for a period of time afterwards. This will provide quantitative information regarding the effect of the intervention. At a one month follow up, these questionnaires will be repeated, and participants will be interviewed about their experiences of the intervention to understand whether there are any issues that need to be considered when using this therapy for SCI patients in hospitals. Using a SCED series design will require us to recruit at least 3 participants.

The information will be analysed to conclude whether it is feasible to use this therapy in this way, and whether it is effective at improving the mental health and quality of life of SCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of a Spinal Cord Injury (SCI)
* Be an inpatient receiving MDT rehabilitation for SCI
* Be able to understand and communicate in English sufficiently to allow for engagement with the intervention, including with the use of reasonable adjustment such as an interpreter, as provided by their usual care team
* Have access to an internet enabled device

Exclusion Criteria:

* Those with a cognitive or physical impairment that would prevent their ability to engage with the intervention

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Recovering Quality of Life-10 (ReQol-10) | Through study completion, approximately 6 weeks
  A measure quality of life (scores range 0 (poor quality of life) - 40 (high quality of life)). Assessed at least three time throughout baseline phase (minimum of one week), at least three times following intervention (minimum of one week) and again at a one month post-intervention follow up
Clinical Outcomes in Routine Evaluation 10 (CORE-10) | through study completion, approximately 6 weeks
  A measure of psychological distress. Scores range from 0 (no/low psychological distress) to 40 (severe psychological distress). To be assessed once at baseline, once following the completion of the intervention and once at a one month post-intervention follow up.
Appraisals of Disability Primary and Secondary Scale-Short Form (ADAPSS-sf) | through study completion, approximately 6 weeks
  A measure to assess cognitive appraisals of, and adjustment to, disability. Scores range from 0-36 with higher scores indicating poorer adjustment. Assessed at least three time throughout baseline phase (minimum of one week), at least three times following intervention (minimum of one week) and again at a one month post-intervention follow up
Comprehensive assessment of Acceptance and Commitment Therapy Processes 10 (CompACT-10) | Through study completion, approximately 6 weeks
  A measure of Psychological flexibility, the core process underlying Acceptance and Commitment Therapy. Higher scores indicate greater psychological flexibility. Assessed at least three time throughout baseline phase (minimum of one week), at least three times following intervention (minimum of one week) and again at a one month post-intervention follow up

SECONDARY OUTCOMES:
Feedback Interview | 1 month post-intervention follow up, approximately week 6
  A qualitative interview conducted with participants to gain information regarding the acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David L Dawson, Principal Investigator — University of Lincoln

IPD SHARING:
Plan to Share IPD: No